CLINICAL TRIAL: NCT03290677
Title: A Phase II Study of Core Needle Biopsy and Cryoablation of an Enlarging Tumor in Patients With Metastatic Lung Cancer and Metastatic Melanoma Receiving Post-progression Immune Checkpoint Inhibitor Therapy
Brief Title: Study of Core Needle Biopsy and Cryoablation of an Enlarging Tumor in Patients With Metastatic Lung Cancer and Metastatic Melanoma Receiving Post-progression Immune Checkpoint Inhibitor Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: William M. Wood Foundation (Unknown)
Responsible Party: Principal Investigator, Meghan Mooradian, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-264
Record Dates: First submitted 2017-09-11; First posted 2017-09-25 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cryosurgery; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-guided Percutaneous Cryoablation of Lung Tumor (Experimental): * Image-guided core needle biopsy to confirm cancer will be perform
  * Patients will undergo cryoablation as a standard procedure
  * cryoablation will be performed with a three-cycle freeze-thaw phase protocol
  * Non-contrast CT images will be obtained in 3 to 5 minutes intervals to visualize the evolving ablation zone
  Interventions: Procedure: Cryoablation; Procedure: Biopsy

INTERVENTIONS:
Procedure: Cryoablation — This involves passing a special needle into the body (cryoprobe) to freeze tumor and kill a small part (not all) of the cancer. The immune system will respond to the damage caused by freezing part of the tumor.
Procedure: Biopsy — Removing a small piece of the affected area to confirm cancer

SUMMARY:
This research study is studying cryoablation (a treatment to kill cancer cells with extreme cold) combined with continued treatment with current immune checkpoint inhibitor as a possible treatment for lung cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved each aspect of this therapy, however this research study is unique because it combines them as a treatment option for the participant's disease. That has not been approved by the FDA.

In this research study, The investigators are...

* Continuing the participant on the participant's immune checkpoint inhibitor therapy even though the participant's doctor believes that the participant's cancer is growing. Since the participant's cancer is growing, there is only a small chance the participant will respond to continued drug therapy.
* Taking a biopsy of the participant's cancer to confirm there is cancer growing in the location to be treated.
* Performing cryoablation on an enlarging tumor. This involves passing a special needle into the participant's body (cryoprobe) to freeze tumor and kill a small part (not all) of the participant's cancer. Your immune system will respond to the damage caused by freezing part of the participant's tumor.
* The investigators are hoping to demonstrate that combining post-progression immune checkpoint inhibitor therapy with cryoablation is safe, and may induce and/or restore an immune response to cancer in other places in the participant's body

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18) with stage IV lung cancer receiving commercial supply immune checkpoint inhibitor therapy with progression of disease, and for whom an additional 4-6 weeks of current therapy (post-progression therapy) is acceptable as standard therapy
* Must have a growing tumor amenable to percutaneous image-guided cryoablation based on routine Interventional Radiology criteria
* Must have measurable disease (by RECIST) independent of the lesion to be ablated. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.

Exclusion Criteria:

* Participants who are receiving an investigational agent(s)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because immune checkpoint inhibitors have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with immune checkpoint inhibitors, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Cumulative Incidence of Treatment Related Serious Adverse Events | 2 years
  The safety and feasibility of the procedure will be determined based on observed adverse events. Cryoablation will be determined safe and feasible to implement in this study population if the cumulative incidence of serious adverse events (SAE) related to cryoablation is no higher than 20%. Adverse events are assessed using Common Terminology Criteria for Adverse Events (CTCAE 4).
Radiologic Response Rate Of Cryoablation | 2 years
  The number of participants that achieve a complete response (CR) or partial response (PR) following cryoablation.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan J Mooradian, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No